CLINICAL TRIAL: NCT03572322
Title: Genetics Tests : How to Improve Management Within Two Medical Specialities
Acronym: ORGAGENE
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: IMT Atlantique Nantes - France (Unknown); Université de Caen Normandie (Other); Université Rennes 1 - France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 35RC17_8819_ORGAGENE
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Genetics; Diagnostic Techniques and Procedures
MeSH Terms: interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Doctors
  Interventions: Other: Focus Group
- Patients
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Focus Group — Focus Group
  Groups: Doctors
Other: Interviews — Interviews
  Groups: Patients

SUMMARY:
This survey will assess discrepancies between official clinical genetics guidelines and practices within 3 West regions of France.

DETAILED DESCRIPTION:
Genetic tests are now widely used in medicine whatever specialities or ages. However genetic tests are not common biological exams as they may either reveal genetic anomalies before any signs (presymptomatic diagnosis) or handle the gene pool of an entire family but not only one patient. Due to these specific managements, genetics tests have required specific laws for nearly 20 years in France.

The French 2011 Bioethics Law (and its decree in 2013) especially issues involving genetic tests now establishes purposes for which genetic data can be disclosed and switch for patient civil responsibility towards his family. This patient has no longer choice and the medical confidentiality might now be breached.

Although specific guidelines practices have been spread by officials, the gap between recommendations and uses tend probably to be huge especially from non-geneticist physicians.

This survey will assess discrepancies between official clinical genetics guidelines and practices within 3 West regions of France.

20 focus groups are intended to be lead with neurologists and oncologists working in hospitals as theses physicians face different genetic issues daily.

20 interviews are scheduled with patients. The investigators aim at collecting information from medical, legal and sociological points of view in order to better understand these gaps.

This will be the first attempt to gather and understand medical practices in the genetic tests area. This could be useful to adapt courses in medical school and along professional life and how to spread them for a deep impact.

ELIGIBILITY:
Inclusion Criteria:

* Specialists in Oncology, Endocrinology, Neurology and Medical Genetics
* Doctors who have already received and returned genetics tests results
* Main hospital exercise (CHU, CH, CRLCC) on the territory of the HUGO interregion regrouping the administrative regions Bretagne, Pays-de-Loire and Centre
* Adults who having benefited genetics tests
* Ability to express oneself easily in French and whose clinical situation allows it

Exclusion Criteria:

* liberal doctor
* Patient refusing to participated in the study
* Medical contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: genetics tests
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Characteristics of the determining factors | through study completion, an average of 1 year
  Characteristics of the determining factors (medical, sociological, ethical and legal) in the medical practices during the implementation of an ECGP

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pasquier, MD, Study Director — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France